CLINICAL TRIAL: NCT05442294
Title: "Juego de Llaves", a Universal School-based Drug Use Prevention Program: A Non-Randomized Control Cluster Trial for the Evaluation of Effectiveness Among Adolescents in Spain (PISUP)
Brief Title: "Juego de LLaves": Study Protocol of a Universal School-based Drug Use Prevention Program (PSIDUP)
Acronym: PSIDUP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Susana Al-Halabí (Other)
Collaborators: United Nations Office on Drugs and Crime (UNODC) (Other Government); Asociación Proyecto Hombre (Unknown)
Responsible Party: Sponsor-Investigator, Susana Al-Halabí, Associate Professor at the Department of Psychology, University of Oviedo
Organization: University of Oviedo (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2021G090 / FUO-22- 023
Record Dates: First submitted 2022-06-15; First posted 2022-07-01 (Actual); Last update posted 2022-07-01 (Actual); Status verified 2022-06

CONDITIONS: Behavior, Addictive; Adolescent - Emotional Problem; Alcohol Abuse; Smoking Behaviors; Adolescent Behavior; Psychological
Keywords: Adolescents; Addictive behaviors; Evaluation; Universal school-based prevention; Transdiagnostic approach
MeSH Terms: conditions — Behavior, Addictive; Alcoholism; Smoking; Adolescent Behavior

STUDY DESIGN:
Intervention Model Description: Non-Randomized Control Cluster Trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Juego de Llaves group (Experimental): This group will receive the prevention program during the academic year in school hours. The prevention program is called Juego de Llaves.
  The main goal of this program is to prevent substance use and engagement in other addictive behaviors. It is intended to be delivered by teachers in a six to twelve session format through different modules that cover the following areas: emotional regulation, cognitive strategies, social interaction, free time, education on drugs and life values
  Interventions: Behavioral: Juego de Llaves
- Control group (No Intervention): The control group will receive the usual teaching activities regarding substance use prevention.

INTERVENTIONS:
Behavioral: Juego de Llaves — The main goal of this program is to prevent substance use and engagement in other addictive behaviors. It is intended to be delivered by teachers in a six to twelve session format through different modules that cover the following areas: emotional regulation, cognitive strategies, social interaction, free time, education on drugs and life values
  Arms: Juego de Llaves group

SUMMARY:
"Juego de Llaves" is a universal school-based drug prevention program for adolescents aged 12-15 years. The outcome evaluation is critical to determine the quality of preventive interventions. This protocol describes the full protocol of the evaluation design, instruments, randomization procedure, follow-ups, and primary outcomes. Method: Non-Randomized Control Cluster Trial in a set of Spanish school centers at the compulsory secondary education level, with follow-ups at 12-, 24- and 36-months. Participants will be allocated to an experimental or control (no intervention) group. Using an electronic ad-hoc designed App, a battery of instruments will be used to assess addictive behaviors, sociodemographic variables, school climate and other transdiagnostic psychological variables. A piloting test will be conducted to test the implementation protocol and to calculate the sample size needed for the outcome evaluation. After implementing the program, longitudinal statistical approaches will be used to inform on the intervention efficacy and potential moderators and mediators. There is a lack of effectiveness assessments of school prevention programs, and it is expected that this protocol will expedite the monitoring and ongoing evaluation in prevention.

ELIGIBILITY:
Inclusion Criteria:

* Schools having secondary education.
* Schools located in Spain.
* Schools willing to participate under the conditions of the study before randomization.

Exclusion Criteria:

* Schools having other interventions with a strong package on substance use prevention targeted the same grades.

Ages: 12 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2500 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2023-06-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Substance use: Tobacco | Past 30-day period
  Ítems from the survey on drug use in secondary education in Spain (ESTUDES) for the National Plan on Drugs
Substance use: Alcohol | Past 30-day period
  Ítems from the survey on drug use in secondary education in Spain (ESTUDES) for the National Plan on Drugs
Substance use: Cannabis | Past 30-day period
  Ítems from the survey on drug use in secondary education in Spain (ESTUDES) for the National Plan on Drugs
Non-substance use behavior: Gaming | Past 30-day period
  Ítems from the survey on drug use in secondary education in Spain (ESTUDES) for the National Plan on Drugs
Non-substance use behavior: Gambling | Past 30-day period
  Ítems from the survey on drug use in secondary education in Spain (ESTUDES) for the National Plan on Drugs
Reinforcement ratio | Past-year period
  Ad-hoc questionnaire (SAUPI; unpublished)
Consecuences of addictive behaviors | Past 30-day period
  ARSS-SUV (adapted from Murphy et al., 2005)

SECONDARY OUTCOMES:
Resilience | Past 30-day period
  The Child and Youth Resilience Measure, CYMR (Resilience Research Centre, 2018)
Behavioral problemas | Past 30-day period
  Strengths and Difficulties Questionnaire (25-item version), SDQ (Ortuño-Sierra et al., 2018)
Emotion regulation | Past 30-day period
  The Emotional Regulation Questionnaire - adolescents, ERQ-CA (Navarro et al., 2018)
Suicidal behavior | Past 30-day period
  The Paykel Suicide Scale, PSS (Fonseca-Pedrero et al., 2018)
Impulsivity | Past 30-day period
  The Scale of Impulsivity for Children and Adolescents BUPPS-P-NA (Caneto et al., 2020)

CONTACTS AND LOCATIONS:
Locations (1):
- Grupo de Conductas Adictivas, University of Oviedo, Oviedo, Principality of Asturias, Spain

REFERENCES:
- See also: Related Info — https://proyectohombre.es/juego-de-llaves-eso/